CLINICAL TRIAL: NCT04183218
Title: Characterizing Chemo-Radiotherapy Treatment-Related Cardiac Changes
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: MC1723; NCI-2019-07938 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1723 (Other: Mayo Clinic in Arizona); 17-008401 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2019-11-27; First posted 2019-12-03 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Clinical Stage 0 Esophageal Adenocarcinoma AJCC V8; Clinical Stage 0 Esophageal Squamous Cell Carcinoma AJCC V8; Clinical Stage I Esophageal Adenocarcinoma AJCC V8; Clinical Stage I Esophageal Squamous Cell Carcinoma AJCC V8; Clinical Stage II Esophageal Adenocarcinoma AJCC V8; Clinical Stage II Esophageal Squamous Cell Carcinoma AJCC V8; Clinical Stage IIA Esophageal Adenocarcinoma AJCC V8; Clinical Stage IIB Esophageal Adenocarcinoma AJCC V8; Clinical Stage III Esophageal Adenocarcinoma AJCC V8; Clinical Stage III Esophageal Squamous Cell Carcinoma AJCC V8; Localized Esophageal Carcinoma; Localized Lung Carcinoma; Pathologic Stage 0 Esophageal Adenocarcinoma AJCC V8; Pathologic Stage 0 Esophageal Squamous Cell Carcinoma AJCC V8; Pathologic Stage I Esophageal Adenocarcinoma AJCC V8; Pathologic Stage I Esophageal Squamous Cell Carcinoma AJCC V8; Pathologic Stage IA Esophageal Adenocarcinoma AJCC V8; Pathologic Stage IA Esophageal Squamous Cell Carcinoma AJCC V8; Pathologic Stage IB Esophageal Adenocarcinoma AJCC V8; Pathologic Stage IB Esophageal Squamous Cell Carcinoma AJCC V8; Pathologic Stage IC Esophageal Adenocarcinoma AJCC V8; Pathologic Stage II Esophageal Adenocarcinoma AJCC V8; Pathologic Stage II Esophageal Squamous Cell Carcinoma AJCC V8; Pathologic Stage IIA Esophageal Adenocarcinoma AJCC V8; Pathologic Stage IIA Esophageal Squamous Cell Carcinoma AJCC V8; Pathologic Stage IIB Esophageal Adenocarcinoma AJCC V8; Pathologic Stage IIB Esophageal Squamous Cell Carcinoma AJCC V8; Pathologic Stage III Esophageal Adenocarcinoma AJCC V8; Pathologic Stage III Esophageal Squamous Cell Carcinoma AJCC V8; Pathologic Stage IIIA Esophageal Adenocarcinoma AJCC V8; Pathologic Stage IIIA Esophageal Squamous Cell Carcinoma AJCC V8; Pathologic Stage IIIB Esophageal Adenocarcinoma AJCC V8; Pathologic Stage IIIB Esophageal Squamous Cell Carcinoma AJCC V8; Postneoadjuvant Therapy Stage I Esophageal Adenocarcinoma AJCC V8; Postneoadjuvant Therapy Stage I Esophageal Squamous Cell Carcinoma AJCC V8; Postneoadjuvant Therapy Stage II Esophageal Adenocarcinoma AJCC V8; Postneoadjuvant Therapy Stage II Esophageal Squamous Cell Carcinoma AJCC V8; Postneoadjuvant Therapy Stage III Esophageal Adenocarcinoma AJCC V8; Postneoadjuvant Therapy Stage III Esophageal Squamous Cell Carcinoma AJCC V8; Postneoadjuvant Therapy Stage IIIA Esophageal Adenocarcinoma AJCC V8; Postneoadjuvant Therapy Stage IIIA Esophageal Squamous Cell Carcinoma AJCC V8; Postneoadjuvant Therapy Stage IIIB Esophageal Adenocarcinoma AJCC V8; Postneoadjuvant Therapy Stage IIIB Esophageal Squamous Cell Carcinoma AJCC V8; Stage 0 Lung Cancer AJCC V8; Stage I Lung Cancer AJCC V8; Stage IA1 Lung Cancer AJCC V8; Stage IA2 Lung Cancer AJCC V8; Stage IA3 Lung Cancer AJCC V8; Stage IB Lung Cancer AJCC V8; Stage II Lung Cancer AJCC V8; Stage IIA Lung Cancer AJCC V8; Stage IIB Lung Cancer AJCC V8; Stage III Lung Cancer AJCC V8; Stage IIIA Lung Cancer AJCC V8; Stage IIIB Lung Cancer AJCC V8; Stage IIIC Lung Cancer AJCC V8
MeSH Terms: conditions — Lung Neoplasms | interventions — Specimen Handling; Chemoradiotherapy; Radiotherapy; Radiation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (cardiac monitoring): Patients receive cardiac monitor implants then undergo standard of care RT or CRT at the discretion of the treating physician. Patients also undergo blood sample collection at baseline, 4 weeks, 3, 9, and 12 months.
  Interventions: Procedure: Biospecimen Collection; Device: Cardiac Event Monitor; Other: Chemoradiotherapy; Radiation: Radiation Therapy

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo biospecimen collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Device: Cardiac Event Monitor — Receive cardiac monitor
Other: Chemoradiotherapy — Undergo CRT
  Other Names: Chemoradiation; CRT; CRTx; Radiochemotherapy; RCTx; RT-CT
Radiation: Radiation Therapy — Undergo RT
  Other Names: Cancer Radiotherapy; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation

SUMMARY:
This trial studies cardiac changes after radiation or chemo-radiation for the treatment of lung or esophageal cancer that has not spread to other places in the body (non-metastatic) or has not come back (non-recurrent). Continuous cardiac monitoring with an implanted device may help to identify cardiac changes that would remain unnoticed, and facilitate the treatment of these early cardiac changes as part of standard care.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the 12-month cardiac event rate after radiation or chemo-radiation for the treatment of lung or esophageal cancer.

EXPLORATORY OBJECTIVES:

I. Define the spectrum of cardiac toxicity among chemoradiotherapy (CRT) patients at highest risk of cardiac toxicity.

II. Establish the timeline of cardiac toxicity development and identify early predictive findings of permanent damage.

III. Characterize the areas of the heart at highest risk for persistent cardiac damage.

IV. Identify a dose response threshold for radiotherapy (RT) damage in different areas of the heart.

V. Improve survival by alerting the cardiology team of the need for life-saving standard of care interventions.

VI. Describe medical interventions employed for the cardiac events identified in the study.

OUTLINE:

Patients receive cardiac monitor implants then undergo standard of care RT or CRT at the discretion of the treating physician. Patients also undergo blood sample collection at baseline, 4 weeks, 3, 9, and 12 months.

After completion of study treatment, patients are followed up at 4 weeks, 3, 9 and 12 months post RT.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Planned standard of care curative thoracic RT or CRT with anticipated heart V40 > 20 cc (At least 20 cc of the heart should receive a dose of 40 gray [Gy] or higher)
* Able to follow-up at all specified standard of care time-points
* Patients can receive treatment as part of the standard of care or in a different study
* Receiving radiation treatment to an area close to the heart, for example gastroesophageal junction cancer, hilar lung cancer, or mainstem bronchus lung cancer
* Any type of systemic therapy or surgery before during or after radiation is acceptable
* Prior radiation to other areas is acceptable
* Planned radiation doses equal or higher than 40 Gy

Exclusion Criteria:

* Metastatic disease
* Recurrent disease
* Patient receiving radiation prescription doses lower than 40 Gy
* No prior radiation that included any part of the heart is acceptable
* No thoracic re-irradiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-metastatic, non-recurrent lung and esophageal cancer patients who are receiving thoracic radiotherapy
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2024-01-06 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
Cardiac event rate at 12 months | Up to 12 months
  Assessed as any cardiac event after registration, including electrophysiological changes as defined by the continuous insertable cardiac monitor (ICM); congestive heart failure (CHF); myocardial infarction; pericarditis or myocarditis; cardiac ablation or cardiac pacemaker; cardiac stent placement or any coronary procedure for coronary damage; or any cardiac event as defined by the patients' medical records or autopsy if done.

SECONDARY OUTCOMES:
Loco-regional recurrence | Up to 12 months
  Loco-regional recurrence is defined as local recurrences of the cancer in the same location where the disease was found on any diagnostic or staging study.
Disease-free survival | Up to 12 months
  Disease- free survival is defined as the time from study registration until any disease recurrence or death.
Distant recurrence | Up to 12 months
  Distant recurrence is defined as metastatic cancer (cancer that has spread to organs or tissues far from the original cancer) that has either been biopsy confirmed or clinically diagnosed as recurrent.
Cardiac event free survival | Up to 12 months
  Cardiac event free survival is defined as the time from registration to any cardiac event or death.
Cardiac death | Up to 12 months
  Cardiac death is defined as the time from registration to death due to cardiac reasons. Cardiac death would include documented congestive heart failure, myocardial infarction, arrhythmia*, heart block*, or any other cardiac cause documented in the medical records, death certificate, or autopsy as one of the major contributing causes of death. *Any lethal electrophysiologic change documented by before death would also be included.
Overall survival | Up to 12 months
  Overall survival is defined as the time from registration to death due to any cause.
Incidence of acute adverse events (AE) | Within the first 6 months from the date of enrollment
  Adverse Event incidence and severity will be measured by the Common Terminology Criteria for Adverse Events (CTCAE) 5.0.
Incidence of late adverse events | After the first 6 months from the date of enrollment
  Adverse Event incidence and severity will be measured by the Common Terminology Criteria for Adverse Events (CTCAE) 5.0.
Cause specific survival | Up to 12 months
  Cause specific survival is defined as the time from registration to death due to cancer.

OTHER OUTCOMES:
Imaging changes | Baseline up to 12 months
  Imaging changes in the heart substructures associated with occurrence of cardiac events will be an exploratory component of this trial. Changes will be described at each time point using frequency distributions.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos E. Vargas, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials